CLINICAL TRIAL: NCT04191473
Title: Comparison of Precutting vs Conventional Endoscopic Mucosal Resection of Intermediate-Size Colorectal Polyps
Brief Title: Comparison of EMR-P With Conventional EMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V2.0
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-12

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group P (Experimental)
  Interventions: Procedure: EMR-P
- group C (Other)
  Interventions: Procedure: CEMR

INTERVENTIONS:
Procedure: EMR-P — After submucosal injection, we use ESD knife or the tip of the entrapment device to loop around the lesion, and then overlapped the loop tangent with the entrapment device. After tightening the entrapment device, all the tumor tissues were confirmed to enter the entrapment device, and the tissues were removed.
  Arms: group P
Procedure: CEMR — A liquid pad was formed by injecting 0.9% normal saline with meilan solution into submucosa,and then overlapped the loop tangent with the entrapment device. After tightening the entrapment device, all the tumor tissues were confirmed to enter the entrapment device, and the tissues were removed.
  Arms: group C

SUMMARY:
Colorectal cancer is the third most common cancer in men and the second most common cancer in women.There are about 14 million cases of colonoscopy in the United States every year. In recent years, the incidence of colorectal cancer in China has risen sharply, becoming a serious threat to people's health.For small(≤ 9mm) lesions, endoscopic biopsy forceps and cold snare polypectomy can be used to remove.For larger lesions, especially laterally spreading tumor,endoscopic mucosal resection is a classic method of treatment.With the increasing diameter of the lesion size(> 20mm),we also need to adopt endoscopic piecemeal mucosal resection or endoscopic submucosal dissection.

As IT, Hook knife, BB, and other devices appear constantly, foreign researchers recently adopted a variation of conventional EMR（CEMR）, namely endoscopic mucosal resection with circumferential precutting(EMR - P).The technology is superior to conventional EMR for 10 to 20 mm polyps.Moreover, preliminary studies suggest that it has good safety and efficacy, and may be a better method for treatment of 10-20mm polyps under colonoscopy.

This clinical trial is being conducted to compare the efficacy and safety of two methods of polypectomy, CEMR and EMR-P, for 10-20mm colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* One polyp or lesion of 10-20mm at the most proximal of colorectal
* Adult patients (≥18 years old)
* Polyps other than pedicled polyps

Exclusion Criteria:

* There was submucosal infiltration under endoscope
* Residual lesions after endoscopic resection
* Inflammatory bowel disease, familial polyps, electrolyte abnormalities, coagulation disorders, or severe organ failure
* Pregnant or nursing
* No informed consent has been signed
* Patients taking NSAIDs or other anticoagulants
* sedated colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 rate | 7 days
  en bloc resection with a histologically confirmed negative resection margin
En bloc rate | immediately
  endoscopically assessed removal of the lesion in one piece

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Renmin Hospital of Yuyao City, Yuyao, Zhejiang